CLINICAL TRIAL: NCT01682668
Title: Role of the Subthalamic Nucleus in the Control of Movement: Physiopathology of Akinesia in Parkinson's Disease.
Brief Title: Subthalamic Nucleus, Akinesia and Parkinson's Disease
Acronym: GB-MOV
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C11-40; 2012-A00225-38 (Registry Identifier: IDRCB)
Record Dates: First submitted 2012-07-19; First posted 2012-09-11 (Estimated); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Parkinson's Disease
Keywords: parkinson's disease; subthalamic nucleus; akinesia; gait initiation; neuronal activity; before STN stimulation; with STN stimulation; functional MRI
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Frequency of subthalamic stimulation (Experimental): Comparison between healthy controls and PD patients (non-operable patients or who will be operated or already operated)
  Interventions: Procedure: Bilateral subthalamic stimulation

INTERVENTIONS:
Procedure: Bilateral subthalamic stimulation

SUMMARY:
This program aims to understand the role of the subthalamic nucleus in the control of the movement in healthy humans and patients with Parkinson's disease, how the STN dysfunction contributes to akinesia and how the STN stimulation improves motor signs in PD patients .

ELIGIBILITY:
Inclusion criteria for patients who will be operated

1. Diagnosis of idiopathic Parkinson's disease (according to the criteria of the United Kingdom Parkinson's Disease Society Brain Bank)
2. Age between 18 and 70;
3. Motor complications in the form of fluctuations in motor state or dyskinesias induced by dopaminergic therapy, despite medical treatment optimum;
4. Other medical conditions that are stable or do not interfere with the procedure proposed;
5. Excellent responsiveness to levodopa (UPDRS motor score improvement greater than 50% in the acute levodopa test)
6. Brain MRI without abnormality
7. Normality of biological examinations
8. Person who has voluntarily and informedly agreed to participate in the study (signature of a written consent)
9. Patient with social health insurance

Criteria for non-inclusion of Parkinsonian patients who will be operated

1. Contraindication to examinations necessary for inclusion
2. Evolutionary psychiatric pathology;
3. Dementia(MMS<24/30);
4. Patients with a medical condition that makes surgery dangerous neuro-surgical;
5. Bleeding-promoting diseases and laboratory test abnormalities clotting;
6. Existence of contraindications to MRI (cardiac or neural pacemaker, clips ferromagnetic surgeries, implants and metal objects, foreign bodies intraocular, pregnancy, claustrophobia).
7. Taking drugs interfering with coagulation for 1 month before intervention.
8. Persons under guardianship, curatorship or any other administrative or judicial measure deprivation of rights and liberty

Selection criteria for non-operated patients

1. Diagnosis of idiopathic Parkinson's disease (according to the criteria of the United Kingdom Parkinson's Disease Society Brain Bank);
2. Age between 18 and 70;
3. Other medical conditions that are stable or do not interfere with the proposed protocol;
4. Presence of axial signs (gait and/or balance disorders) no improved by antiparkinsonian treatment
5. Brain MRI without notable abnormality
6. Normality of biological examinations
7. Person who has voluntarily and informedly agreed to participate in the study (signature of a written consent)
8. Patient with social health insurance

Criteria for non-inclusion of non-operated patients

1. Contraindication to examinations necessary for inclusion
2. Progressive psychiatric pathology;
3. Dementia (MMS<24/30);
4. Existence of contraindications to MRI (cardiac or neural pacemaker, clips ferromagnetic surgeries, implants and metal objects, foreign bodies intraocular, pregnancy, claustrophobia).
5. Persons under guardianship, curatorship or any other administrative or judicial measuredeprivation of rights and liberty

Inclusion criteria for group 3 patients (already operated)

1. Diagnosis of idiopathic Parkinson's disease (according to the criteria of the United Kingdom Parkinson's Disease Society Brain Bank);
2. Bilateral deep brain stimulation of the subthalamic nucleus for more than 1 year
3. Age between 18 and 70;
4. Person who has voluntarily and informedly agreed to participate in the study (signature of a written consent)
5. Patient with social health insurance

Criteria for non-inclusion of Parkinsonian patients (already operated)

1. Contraindication to examinations necessary for inclusion
2. Evolutionary psychiatric pathology;
3. Dementia(MMS<24/30);
4. Persons under guardianship, curatorship or any other administrative or judicial measure deprivation of rights and liberty

Inclusion criteria for healthy subjects

1. Age between 18 and 70 years old
2. Normal neurological examination
3. Person who voluntarily and informedly agreed to participate in the study (signature of a written consent)
4. Patient with social health insurance

Criteria for non-inclusion of healthy subjects

1. Persons under guardianship, curatorship or any other administrative or judicial measure of deprivation of rights and freedom
2. Existence of neurological, orthopedic or psychiatric history
3. Existence of contraindications to MRI (cardiac or neural pacemaker, ferromagnetic surgical clips, implants and metallic objects, foreign bodies intraocular, pregnancy, claustrophobia).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2013-02 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Firing rate of the subthalamic neurons | During surgery for bilateral STN stimulation
  Changes in the neuronal activity of the STN before, during and after the execution of an arm movement

SECONDARY OUTCOMES:
Evoked related potentials of the STN | 3-5 days after surgery for bilateral STN stimulation
  Local-field potentials recordings with DBS electrodes when performing the execution of an arm movement or gait initiation
Biomechanical parameters of gait initiation | 6 months
  Gait initiation parameters by using a forceplate and EMG recordings

OTHER OUTCOMES:
BOLD signal during fMRI | 1 month before surgery
  Changes in the BOLD signal during fMRI with virtual imagery of movement
real-life assessment | 1 month after surgery
  recording using the percept device

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Laure Welter, MD, PhD, Principal Investigator — GHPS, APHP, Paris, France
Locations (2):
- France (2):
  - CIC-GHPS, Paris
  - Groupe Hospitalier Pitie-Salpêtrière, Paris